CLINICAL TRIAL: NCT03011099
Title: Improving Gait Performance in Individuals With Spinal Cord Injuries: an Intervention Using Robotic Exoskeletons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Matthew Edward Davis, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-13-0536
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic exoskeleton training (Experimental): During the training, subjects will wear a lower extremity exoskeleton robotic walking device. Subjects will participate in individualized treatment sessions which may include: sit to stand, static and dynamic standing balance, weight shifting, walking, turning, and stand to sit. Each training session will last up to 90 minutes (60 minutes of training with 30 minutes for setup, don/doff of device) and training will be held 5 days per week for 3 weeks with a total of 15 sessions. During the training period, subjects will be required to maintain the same amount and level of regular daily physical activity and exercise.
  Interventions: Device: Robotic exoskeleton training
- Conventional Physical Therapy (Active Comparator): During the training, subjects will receive conventional physical therapy that is designed to facilitate/promote gait. This will include individualized treatment sessions for each subject and may involve stretching, strengthening, balance training, standing, and gait training. Subjects will not be able to participate in any form of robotic assisted or body weight supported treadmill training. Each training session will last up to 60 minutes and training will be held 5 days per week for 3 weeks with a total of 15 sessions. Consistent with the RET group, subjects will be required to maintain the same amount and level of regular daily physical activity and exercise during study period.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Device: Robotic exoskeleton training — During the training, subjects will wear a lower extremity exoskeleton robotic walking device. Subjects will participate in individualized treatment sessions which may include: sit to stand, static and dynamic standing balance, weight shifting, walking, turning, and stand to sit. Each training session will last up to 90 minutes (60 minutes of training with 30 minutes for setup, don/doff of device) and training will be held 5 days per week for 3 weeks with a total of 15 sessions. During the training period, subjects will be required to maintain the same amount and level of regular daily physical activity and exercise.
  Arms: Robotic exoskeleton training
Other: Conventional physical therapy — During the training, subjects will receive conventional physical therapy that is designed to facilitate/promote gait. This will include individualized treatment sessions for each subject and may involve stretching, strengthening, balance training, standing, and gait training. Subjects will not be able to participate in any form of robotic assisted or body weight supported treadmill training. Each training session will last up to 60 minutes and training will be held 5 days per week for 3 weeks with a total of 15 sessions. Consistent with the RET group, subjects will be required to maintain the same amount and level of regular daily physical activity and exercise during study period.
  Arms: Conventional Physical Therapy

SUMMARY:
The purpose of this study is to investigate whether robotic exoskeleton training can improve walking performance after SCI as compared to conventional physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Motor Incomplete spinal cord injury, as classified by American Spinal Injury Association guidelines, above the lumbar level (T12 and above).
* Able to independently stand for two minutes with or without an assistive device and with or without orthoses distal to the knee.
* Male or non-pregnant woman
* ≥ 18-years of age
* At least 6 months after injury
* Height between 5'2" and 6'2" (150-188 cm)
* Weight ≤ 220 pounds (100 kg)
* Ability to perform informed consent

Exclusion Criteria:

* Presence of clinical signs of lower motor neuron injury
* History of severe neurologic injuries other than SCI (MS, CP, ALS, TBI, CVA, etc.)
* Severe comorbidities: active infections, heart, lung, or circulatory conditions, pressure ulcers.
* Documented severe osteoporosis affecting the hip and spine
* Severe spasticity in the lower extremities (Modified Ashworth ≥ 3) or uncontrolled clonus
* Unstable spine
* Unhealed limb or pelvic fractures
* Skin issues that would prevent wearing the device
* Range of motion restrictions that would prevent subject from achieving a normal, reciprocal gait pattern, or would restrict a subject from completing normal sit to stand or stand to sit transitions.
* Upper extremity strength deficits that limit ability to balance with a front rolling walker or crutches.
* Heterotopic ossification that resists functional range of motion in lower extremities
* Contractures (>15 degrees at the hips or >20 degrees at the knees)
* Psychiatric or cognitive comorbidities resulting in motor planning or impulsivity concerns
* Colostomy
* Have received any physical therapy intervention within 3 months prior to enrolment in the study
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Chang SH, Afzal T; TIRR SCI Clinical Exoskeleton Group; Berliner J, Francisco GE. Exoskeleton-assisted gait training to improve gait in individuals with spinal cord injury: a pilot randomized study. Pilot Feasibility Stud. 2018 Mar 5;4:62. doi: 10.1186/s40814-018-0247-y. eCollection 2018. PMID 29556414

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant dropped out of the study after signing the consent before randomization.
Period: Overall Study
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy
Started | 6 | 5
Completed | 6 | 3
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Over Ground Gait Speed as Assessed by the 10 Meter Walk Test
Description: The 10 Meter Walk Test assesses the time taken to walk 10 meters.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy
Number analyzed (Participants) | 6 | 3
seconds | -6.815 (9.58) | -0.5 (4.02)

2. Primary Outcome: Change in Walking Endurance as Assessed by the 6 Minute Walk Test
Description: The 6 Minute Walk Test assesses the distance walked in 6 minutes.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: feet
Groups:
- Robotic Exoskeleton Training: Robotic exoskeleton training: During the training, subjects will wear a lower extremity exoskeleton robotic walking device. Subjects will participate in individualized treatment sessions which may include: sit to stand, static and dynamic standing balance, weight shifting, walking, turning, and stand to sit. Each training session will last up to 90 minutes
- Conventional Physical Therapy: Conventional physical therapy: During the training, subjects will receive conventional physical therapy that is designed to facilitate/promote gait. This will include individualized treatment sessions for each subject and may involve stretching, strengthening, balance training, standing, and gait training
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy
Number analyzed (Participants) | 6 | 3
feet | 34.3833 (42.83) | 25.3 (25.96)

3. Primary Outcome: Change in Dynamic Mobility Assessment as Determined by the Timed Up and Go Test
Description: The Timed Up and Go test assessed the time it takes to stand from a sitting position, complete a 3 meter walk, and then return to sitting.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: Second
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy
Number analyzed (Participants) | 6 | 3
Second | -10.575 (17.31) | -1.59 (0.44)

4. Primary Outcome: Change in Muscle Activity as Assessed by Surface Electromyography (EMG)
Description: Surface EMG sensors will be placed on the skin of subjects' lower extremities and trunk to measure muscle activity. Only one participant data was analyzed. Emg was recorded from the soleus, gastrocnemius, tibialis anterior, rectus femoris, vastus medialis, bicep femoris and semitendinosus muscles. The outcome measure is the %age change between the baseline and 4 week assessments. Negative values denotes decrease in muscle activity at 4 week compared to baseline.
Time Frame: baseline, week 4
Population: This measure was later added to the protocol and hence data was collected from one participant only.
Measure: Number; unit: percentage of muscle activity change
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy
Number analyzed (Participants) | 1 | 0
percentage of muscle activity change
  Change in soleus activity | -44 |
  Change in gastrocnemius activity | -37 |
  Change in tibialis anterior activity | 57 |
  Change in Rectus Femoris activity | 12 |
  Change in Vastus Medialis activity | -18 |
  Change in Bicep Femoris activity | 33 |
  Change in Semitendinosus activity | 32 |

5. Primary Outcome: Change in Energy Expenditure During Walking as Assessed by Oxygen Cost
Description: Oxygen cost will be calculated from oxygen consumption as the product of gait speed and body weight.20 Oxygen consumption will be calculated on a breath-by-breath basis measured by a portable metabolic system (Cosmed K4b2).
Time Frame: baseline, week 4
Population: The metabolic expenditure was only measured for two subjects who completed the Robotic exoskeleton training at the end of the study. The equipment to use metabolic expenditure was not available at that time of enrollment of the population at the beginning of the study. Therefore data was only collected once the equipment became operational.
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy
Number analyzed (Participants) | 2 | 0
ml/min/kg | -0.84 (0.56) |

6. Secondary Outcome: Change in Gait Characteristics as Assessed by the GAITRite Walkway (Cadence)
Description: Gait quality will be measured with the GAITRite Walkway which can quantify step cadence, step length, step time, double support time, and symmetry. Cadence is measured as steps/min. Change in cadence is reported as difference between baseline and post assessment.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy
Number analyzed (Participants) | 6 | 3
steps/min | 0.12 (0.17) | 0.08 (0.11)

7. Secondary Outcome: Change in Gait Characteristics as Assessed by the GAITRite Walkway (Step Length)
Description: Gait quality will be measured with the GAITRite Walkway which can quantify step cadence, step length, step time, double support time, and symmetry. The change in step length between baseline and post assessment is reported. Negative value denotes decrease in step length.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy
Number analyzed (Participants) | 6 | 3
cm | 0.04 (0.11) | -0.03 (0.08)

8. Secondary Outcome: Change in Gait Characteristics as Assessed by the GAITRite Walkway (Step Time)
Description: Gait quality will be measured with the GAITRite Walkway which can quantify step cadence, step length, step time, double support time, and symmetry. The outcome measure is the difference in step time between pre and post assessment. Negative value denotes decrease in step time (implying faster step time at post).
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy
Number analyzed (Participants) | 6 | 3
seconds | -0.09 (0.13) | -0.02 (0.11)

9. Secondary Outcome: Change in Lower Extremity Strength as Assessed by American Spinal Injury Association (ASIA) Lower Extremity Motor Score (LEMS)
Description: The ASIA (American Spinal Injury Association) assessment protocol consists of two sensory examinations, a motor examination and a classification framework (the impairment scale) to quantify the severity of the spinal cord injury. The scale informs about the functionality of the patient. The range of scores is 0 to 5, and high values represent better outcome. Following is the description of the range:
  0 = total paralysis
  1. = palpable or visible contraction
  2. = active movement, full range of motion (ROM) with gravity eliminated
  3. = active movement, full ROM against gravity
  4. = active movement, full ROM against gravity and moderate resistance in a muscle specific position
  5. = (normal) active movement, full ROM against gravity and full resistance in a functional muscle position expected from an otherwise unimpaired person
  We report the difference between baseline and 4week assessments. Negative value denotes decrease at post assessment.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy
Number analyzed (Participants) | 6 | 3
units on a scale | 0.42 (2.15) | -0.17 (0.41)

10. Secondary Outcome: Exoskeleton User Feedback as Assessed by a Questionnaire
Description: A questionnaire will be administered to allow participants to provide feedback regarding their experiences during training sessions with the exoskeleton. The units on a scale was used to measure the feedback. The range of the scale was 1-5. '1' refers to very satisfied and '5' refers to very dissatisfied. '1' refers to a better outcome.
Time Frame: week 4
Population: This measure was only recorded from the participants in the robotic exoskeleton training group. This outcome was mainly related to the feedback of the participants after using the exoskeleton at the end of the training.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy
Number analyzed (Participants) | 6 | 0
units on a scale | 1.83 (0.75) |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant during their participation in the study. the study protocol was 1 month long.
Arm/Group | Robotic Exoskeleton Training | Conventional Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 1/6 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Exoskeleton Training (N=6) | Conventional Physical Therapy (N=3)
swelling and pain in foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes